CLINICAL TRIAL: NCT02525848
Title: Aprepitant Versus Gabapentin Prophylaxis for Postoperative Nausea and Vomiting in Laparoscopic Gynecological Surgeries
Acronym: PONV
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, MD, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00008718/ reference no. 104
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone; Calcium Dobesilate; Gabapentin; Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- dexamethasone (Active Comparator): intravenous dexamethasone 8 mg 2 minutes before induction of anesthesia;
  Interventions: Drug: dexamethasone
- gapabentin (Active Comparator): oral gabapentin 600 mg 1 hour before induction of anesthesia
  Interventions: Drug: dexamethasone; Drug: Gabapentin
- Aprepitant (Active Comparator): aprepitan 80mg 1 hour before induction of anesthesia.
  Interventions: Drug: dexamethasone; Drug: Aprepitant

INTERVENTIONS:
Drug: dexamethasone — dexamethasone 8 mg iv 2 minutes before induction of anesthesia
  Other Names: Decadron
Drug: Gabapentin — oral gabapentin 600 mg 1 hour before induction of anesthesia
  Other Names: Neurontin
  Arms: gapabentin
Drug: Aprepitant — oral aprepitan 80mg 1 hour before induction of anesthesia.
  Other Names: Emend
  Arms: Aprepitant

SUMMARY:
To evaluate the efficacy of pre-empetive administration of Aprepitant, Versus Gabapentin prophylaxis for reducing the incidence of postoperative nausea and vomiting in Laproscopic gynacological surgeries.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is frequently encountered in the surgical recovery room. Laparoscopic surgery is one important risk factor for increased incidence of PONV. Gabapentin, an anticonvulsant with known postoperative analgesic properties, has shown some activity against PONV. Results from clinical trials evaluating the anti-emetic efficacy of gabapentin are conflicting.

Aprepitant, a neurokinin-1 (NK1) receptor antagonist, blockades the central effects of substance P. Substance P is a neurotransmitter found in central areas associated with emesis such as the dorsal vagal complex and area postrema.

ELIGIBILITY:
Inclusion Criteria:

• ASA physical status I and II aged between 18 and 45 yrs. They undergo Laproscopic gynacological surgeries under general anesthesia.

Exclusion Criteria:

* Central or peripheral neurological pathologies.
* History of drug abuse, chronic pain, or psychiatric disorders.
* Pregnant women
* Patients who took sedatives, antiemetics, or antipruritics within 24 hrs of operation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
incidence (%) of postoperative nausea and vomiting | 24 hours postoperative
  The incidence (%) of PONV will be recorded each 6 hours until 24 hours after discharge from the PACU.

SECONDARY OUTCOMES:
non invasive blood pressure | intra-operative from induction of general anesthesia till end of surgery.
  Noninvasive blood pressure measured immediately after induction of anesthesia ,15 min.30 min.45 min. and 60 min till the end of surgery
heart rate | Intra-operative from induction of anesthesia till end of surgery.
  heart rate recorded immediately after induction of anesthesia ,15 min.30 min.45 min. and 60 min till the end of surgery
side effects | 24 h postoperative.
  Side effects of given drugs will be treated and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assisstant professor in Anesthesia and intensive care department, faculty of medicine, Assiut university, Egypt
Locations (1):
- Hala saad Abdel-Ghaffar, Asyut, Assiut Governorate, Egypt